CLINICAL TRIAL: NCT07051226
Title: Deep Learning-Based Confocal Laser Microendoscopy Feature Atlas Construction and Its Application in Intelligent Diagnosis of Irritable Bowel Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Kaijun Liu, MD, Ph.D,Associate Professor, Associate Chief Physician, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: Ratification NO:2025(203)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Tissue sections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control group
- IBS test group

SUMMARY:
In this study, the healthy control group and IBS patients are taken as the research subjects, and CLE is applied to image and analyze the enrolled persons respectively, to derive and compare the characteristic microstructural images of the healthy control group with those of the IBS patients, to establish a diagnostic model of IBS by using deep learning and to evaluate the diagnostic efficacy of the model for IBS.Participants will undergo colonoscopy and confocal laser microendoscopy, and IBS patients will undergo targeted biopsy in CLE to observe suspicious lesions and lesion margins, and specimens will undergo HE staining and immunohistochemistry testing.

Translated with DeepL.com (free version)

DETAILED DESCRIPTION:
The study is prospective, observational, and diagnostic.

Research methodology Equipment Consumables The equipment consumables used include a colonoscopy operating system, pCLE system, fluorescein sodium injection, and single-use endoscopic biopsy forceps.

Phase 1 Endoscopy All enrolled person receive fluorescein sodium allergy test before pCLE examination, and fluorescein sodium is injected intravenously after observing no allergic reactions such as dizziness, rash, itching, shock, etc. for 15 min. 30 s later, the pCLE probe is placed from the biopsy clamp channel of enteroscopy, and six different intestinal segments of the cecum, ascending colon, transverse colon, descending colon, sigmoid colon, and rectum are examined in order and the images are collected, and each intestinal segment of the pCLE of all person is recorded continuously with 3-minute video recordings (operation is kept within 30 min after the procedure). and more than 4000 images are recorded for each person. During the operation, the probe is gently placed on the mucosal surface and kept as perpendicular to the bowel wall as possible, and the movements are gentle, slow, and soft to avoid mucosal injury. The endoscopist is performing targeted biopsies of all suspicious lesions and lesion margins observed in pCLE.

Pathological analysis After the specimens are fixed in formalin solution and embedded in paraffin, 2 sections with a thickness of 4 μm are cut. The first section is stained with HE to evaluate the mild inflammation of the intestine; the second section is stained with immunohistochemistry to evaluate the mast cell markers and tight junction proteins in the intestinal wall.

Screening of characteristic pCLE images All videos are measured and analyzed by the same experienced endoscopist, after screening all images with good stability, no artifacts, and clear display of microstructures. pCLE images are characterized by a ruler of 10 μm in length in the lower left corner, which allows real-time evaluation of a number of parameters in real time during the operation. Image J image analysis software is used to measure capillary diameter (CD), cell spacing (CS), gland spacing (GS), gland area (GA), and whether sodium fluorescein leak into the crypt lumen in the pCLE field of view. and other indicators. The images are categorized according to the healthy control group and the IBS patient group, and the characteristic images of each group are formed.

Phase 2 Diagnostic model construction of IBS patient images Deep learning is performed based on two sets of characteristic images to construct a diagnostic model for IBS.

Model evaluation Patients with healthy, IBS, early IBD, or celiac disease (total sample size of 30 cases for total diagnostic model efficacy validation in phases 2 and 3) are examined for pCLE in the same way as in phase 1, and high-quality images are screened for discriminative diagnosis of this model and evaluated for accuracy and inter-evaluator agreement of their diagnostic findings.

Phase 3 Construction of a multimodal diagnostic model for images of IBS patients with joint text On the basis of phase 2, the text data of various indicators corresponding to the images are added for joint deep learning to construct a multimodal diagnostic model for IBS patients.

Model evaluation Patients with healthy, IBS, early IBD, or celiac disease (total sample size of 30 cases for validation of diagnostic model efficacy in phases 2 and 3 combined) are examined for pCLE in the same way as in phase 1, with high-quality images and various types of indicators screened for discriminatory diagnosis of this model and evaluated for the accuracy of the diagnostic results and inter-appraisal agreement.

ELIGIBILITY:
Inclusion Criteria:

* ①Healthy control group and test group of IBS with clear clinical diagnosis (Rome IV diagnostic criteria). Healthy controls are free of gastrointestinal symptoms, test results (blood count, CRP, ESR, etc.) and colonoscopy abnormalities.Patients with IBS have recurrent abdominal pain (≥1 day per week on average in the past 3 months), with onset ≥6 months before diagnosis, and the abdominal pain is accompanied by at least two of the following three symptoms: pain related to defecation, change in stool frequency, and change in the shape (appearance) of the feces, and other organic or metabolic disorders are excluded.② Age: between 18 and 80 years old.③ Probe-based confocal Laser Endomicroscopy (pCLE) is required, and patients have good compliance. ④ Normal coagulation function, and biopsies can be obtained for pathological examination.⑤ Voluntary signing of informed consent.

Exclusion Criteria:

* Fluorescein sodium allergy. ②Contraindications to colonoscopy (pregnant or breastfeeding patients, uncooperative psychiatric patients with severe mental disorders, colonic obstruction) or inadequate bowel preparation (Boston Bowel Preparedness Scale score of <2 for any colonic segment).③ Comorbidities with major organ dysfunction (with severe cardiopulmonary disease) or impaired renal function (blood creatinine >450umol/L). ④ Other conditions that, in the judgment of the investigator, make it unsuitable for participation in the study (inflammatory bowel disease, infected IBS, having taken nonsteroidal anti inflammatory drugs, corticosteroids or antibiotics within the last year, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy control group and test group of IBS with clear clinical diagnosis (Rome IV diagnostic criteria). Healthy controls are free of gastrointestinal symptoms, test results (blood count, CRP, ESR, etc.) and colonoscopy abnormalities.Patients with IBS have recurrent abdominal pain (≥1 day per week on average in the past 3 months), with onset ≥6 months before diagnosis, and the abdominal pain is accompanied by at least two of the following three symptoms: pain related to defecation, change in stool frequency, and change in the shape (appearance) of the feces, and other organic or metabolic disorders are excluded.Between the ages of 18 and 80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the accuracy and inter-evaluator agreement of the constructed IBS diagnostic model with the diagnostic results of the Rome IV criteria. | Approximately 15 months from completion of image collection, analysis, deep learning and construction of IBS diagnostic model to validation of diagnostic model performance.
  Diagnostic model constructed from CLE-based image data and multimodal model constructed from fused image joint text data

REFERENCES:
- [Background] Fritscher-Ravens A, Pflaum T, Mosinger M, Ruchay Z, Rocken C, Milla PJ, Das M, Bottner M, Wedel T, Schuppan D. Many Patients With Irritable Bowel Syndrome Have Atypical Food Allergies Not Associated With Immunoglobulin E. Gastroenterology. 2019 Jul;157(1):109-118.e5. doi: 10.1053/j.gastro.2019.03.046. Epub 2019 May 15. PMID 31100380
- [Background] Fritscher-Ravens A, Schuppan D, Ellrichmann M, Schoch S, Rocken C, Brasch J, Bethge J, Bottner M, Klose J, Milla PJ. Confocal endomicroscopy shows food-associated changes in the intestinal mucosa of patients with irritable bowel syndrome. Gastroenterology. 2014 Nov;147(5):1012-20.e4. doi: 10.1053/j.gastro.2014.07.046. Epub 2014 Jul 30. PMID 25083606
- [Background] Bertiaux-Vandaele N, Youmba SB, Belmonte L, Lecleire S, Antonietti M, Gourcerol G, Leroi AM, Dechelotte P, Menard JF, Ducrotte P, Coeffier M. The expression and the cellular distribution of the tight junction proteins are altered in irritable bowel syndrome patients with differences according to the disease subtype. Am J Gastroenterol. 2011 Dec;106(12):2165-73. doi: 10.1038/ajg.2011.257. Epub 2011 Oct 18. PMID 22008894
- [Background] Liu JJ, Rudzinski JK, Mah SJ, Thiesen AL, Bao H, Wine E, Ogg SC, Boulanger P, Fedorak RN, Madsen KL. Epithelial gaps in a rodent model of inflammatory bowel disease: a quantitative validation study. Clin Transl Gastroenterol. 2011 Jun 9;2(6):e3. doi: 10.1038/ctg.2011.2. PMID 23237881
- [Background] Robles-Medranda C, Oleas R, Valero M, Puga-Tejada M, Soria-Alcivar M, Ospina J, Alvarado-Escobar H, Munoz-Jurado G, Baquerizo-Burgos J, Pitanga-Lukashok H. Confocal laser endomicroscopy detects colonic inflammation in patients with irritable bowel syndrome: a prospective study. Endosc Int Open. 2020 Apr;8(4):E550-E557. doi: 10.1055/a-1119-6327. Epub 2020 Mar 23. PMID 32258379
- [Background] Kiesslich R, Goetz M, Angus EM, Hu Q, Guan Y, Potten C, Allen T, Neurath MF, Shroyer NF, Montrose MH, Watson AJ. Identification of epithelial gaps in human small and large intestine by confocal endomicroscopy. Gastroenterology. 2007 Dec;133(6):1769-78. doi: 10.1053/j.gastro.2007.09.011. Epub 2007 Sep 16. PMID 18054549
- [Background] Liu JJ, Wong K, Thiesen AL, Mah SJ, Dieleman LA, Claggett B, Saltzman JR, Fedorak RN. Increased epithelial gaps in the small intestines of patients with inflammatory bowel disease: density matters. Gastrointest Endosc. 2011 Jun;73(6):1174-80. doi: 10.1016/j.gie.2011.01.018. Epub 2011 Mar 11. PMID 21396639
- [Background] ASGE Technology Committee. Confocal laser endomicroscopy. Gastrointest Endosc. 2014 Dec;80(6):928-38. doi: 10.1016/j.gie.2014.06.021. No abstract available. PMID 25442092
- [Background] Piche T, Barbara G, Aubert P, Bruley des Varannes S, Dainese R, Nano JL, Cremon C, Stanghellini V, De Giorgio R, Galmiche JP, Neunlist M. Impaired intestinal barrier integrity in the colon of patients with irritable bowel syndrome: involvement of soluble mediators. Gut. 2009 Feb;58(2):196-201. doi: 10.1136/gut.2007.140806. Epub 2008 Sep 29. PMID 18824556
- [Background] Martinez C, Lobo B, Pigrau M, Ramos L, Gonzalez-Castro AM, Alonso C, Guilarte M, Guila M, de Torres I, Azpiroz F, Santos J, Vicario M. Diarrhoea-predominant irritable bowel syndrome: an organic disorder with structural abnormalities in the jejunal epithelial barrier. Gut. 2013 Aug;62(8):1160-8. doi: 10.1136/gutjnl-2012-302093. Epub 2012 May 25. PMID 22637702
- [Background] Hughes PA, Harrington AM, Castro J, Liebregts T, Adam B, Grasby DJ, Isaacs NJ, Maldeniya L, Martin CM, Persson J, Andrews JM, Holtmann G, Blackshaw LA, Brierley SM. Sensory neuro-immune interactions differ between irritable bowel syndrome subtypes. Gut. 2013 Oct;62(10):1456-65. doi: 10.1136/gutjnl-2011-301856. Epub 2012 Jul 5. PMID 22767422
- [Background] Liu Y, Zhang L, Wang X, Wang Z, Zhang J, Jiang R, Wang X, Wang K, Liu Z, Xia Z, Xu Z, Nie Y, Lv X, Wu X, Zhu H, Duan L. Similar Fecal Microbiota Signatures in Patients With Diarrhea-Predominant Irritable Bowel Syndrome and Patients With Depression. Clin Gastroenterol Hepatol. 2016 Nov;14(11):1602-1611.e5. doi: 10.1016/j.cgh.2016.05.033. Epub 2016 Jun 4. PMID 27266978
- [Background] Martinez C, Gonzalez-Castro A, Vicario M, Santos J. Cellular and molecular basis of intestinal barrier dysfunction in the irritable bowel syndrome. Gut Liver. 2012 Jul;6(3):305-15. doi: 10.5009/gnl.2012.6.3.305. Epub 2012 Jul 12. PMID 22844557
- [Background] Montrose MH. The future of GI and liver research: editorial perspectives: I. Visions of epithelial research. Am J Physiol Gastrointest Liver Physiol. 2003 Apr;284(4):G547-50. doi: 10.1152/ajpgi.00547.2002. PMID 12631555
- [Background] Clayburgh DR, Shen L, Turner JR. A porous defense: the leaky epithelial barrier in intestinal disease. Lab Invest. 2004 Mar;84(3):282-91. doi: 10.1038/labinvest.3700050. PMID 14767487
- [Background] Turcotte JF, Kao D, Mah SJ, Claggett B, Saltzman JR, Fedorak RN, Liu JJ. Breaks in the wall: increased gaps in the intestinal epithelium of irritable bowel syndrome patients identified by confocal laser endomicroscopy (with videos). Gastrointest Endosc. 2013 Apr;77(4):624-30. doi: 10.1016/j.gie.2012.11.006. Epub 2013 Jan 26. PMID 23357497
- [Background] Choghakhori R, Abbasnezhad A, Hasanvand A, Amani R. Inflammatory cytokines and oxidative stress biomarkers in irritable bowel syndrome: Association with digestive symptoms and quality of life. Cytokine. 2017 May;93:34-43. doi: 10.1016/j.cyto.2017.05.005. Epub 2017 May 12. PMID 28506572
- [Background] Bashashati M, Moossavi S, Cremon C, Barbaro MR, Moraveji S, Talmon G, Rezaei N, Hughes PA, Bian ZX, Choi CH, Lee OY, Coeffier M, Chang L, Ohman L, Schmulson MJ, McCallum RW, Simren M, Sharkey KA, Barbara G. Colonic immune cells in irritable bowel syndrome: A systematic review and meta-analysis. Neurogastroenterol Motil. 2018 Jan;30(1). doi: 10.1111/nmo.13192. Epub 2017 Aug 29. PMID 28851005
- [Background] Spiegel BM, Farid M, Esrailian E, Talley J, Chang L. Is irritable bowel syndrome a diagnosis of exclusion?: a survey of primary care providers, gastroenterologists, and IBS experts. Am J Gastroenterol. 2010 Apr;105(4):848-58. doi: 10.1038/ajg.2010.47. Epub 2010 Mar 2. PMID 20197761
- [Background] Begtrup LM, Engsbro AL, Kjeldsen J, Larsen PV, Schaffalitzky de Muckadell O, Bytzer P, Jarbol DE. A positive diagnostic strategy is noninferior to a strategy of exclusion for patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2013 Aug;11(8):956-62.e1. doi: 10.1016/j.cgh.2012.12.038. Epub 2013 Jan 26. PMID 23357491
- [Background] Camilleri M, Halawi H, Oduyebo I. Biomarkers as a diagnostic tool for irritable bowel syndrome: where are we? Expert Rev Gastroenterol Hepatol. 2017 Apr;11(4):303-316. doi: 10.1080/17474124.2017.1288096. Epub 2017 Feb 13. PMID 28128666
- [Background] Nakov R, Snegarova V, Dimitrova-Yurukova D, Velikova T. Biomarkers in Irritable Bowel Syndrome: Biological Rationale and Diagnostic Value. Dig Dis. 2022;40(1):23-32. doi: 10.1159/000516027. Epub 2021 Mar 22. PMID 33752201
- [Background] Ford AC, Lacy BE, Talley NJ. Irritable Bowel Syndrome. N Engl J Med. 2017 Jun 29;376(26):2566-2578. doi: 10.1056/NEJMra1607547. No abstract available. PMID 28657875
- [Background] Saha L. Irritable bowel syndrome: pathogenesis, diagnosis, treatment, and evidence-based medicine. World J Gastroenterol. 2014 Jun 14;20(22):6759-73. doi: 10.3748/wjg.v20.i22.6759. PMID 24944467
- [Background] Chey WD, Kurlander J, Eswaran S. Irritable bowel syndrome: a clinical review. JAMA. 2015 Mar 3;313(9):949-58. doi: 10.1001/jama.2015.0954. PMID 25734736
- [Background] Buono JL, Mathur K, Averitt AJ, Andrae DA. Economic burden of inadequate symptom control among US commercially insured patients with irritable bowel syndrome with diarrhea. J Med Econ. 2017 Apr;20(4):353-362. doi: 10.1080/13696998.2016.1269016. Epub 2017 Jan 4. PMID 27919177
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Choi MG, Jung HK. Health related quality of life in functional gastrointestinal disorders in Asia. J Neurogastroenterol Motil. 2011 Jul;17(3):245-51. doi: 10.5056/jnm.2011.17.3.245. Epub 2011 Jul 13. PMID 21860816
- [Background] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Background] Sood R, Law GR, Ford AC. Diagnosis of IBS: symptoms, symptom-based criteria, biomarkers or 'psychomarkers'? Nat Rev Gastroenterol Hepatol. 2014 Nov;11(11):683-91. doi: 10.1038/nrgastro.2014.127. Epub 2014 Jul 29. PMID 25069544
- [Background] Camilleri M. Diagnosis and Treatment of Irritable Bowel Syndrome: A Review. JAMA. 2021 Mar 2;325(9):865-877. doi: 10.1001/jama.2020.22532. PMID 33651094
- [Background] Ford AC, Sperber AD, Corsetti M, Camilleri M. Irritable bowel syndrome. Lancet. 2020 Nov 21;396(10263):1675-1688. doi: 10.1016/S0140-6736(20)31548-8. Epub 2020 Oct 10. PMID 33049223